CLINICAL TRIAL: NCT05404789
Title: Tolerance of Centrifuge-induced Acceleration in Subjects With Diabetes Mellitus and Cardiac Arrhythmia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: Civil Aerospace Medical Institute (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 21-0078
Record Dates: First submitted 2021-08-26; First posted 2022-06-03 (Actual); Last update posted 2022-11-04 (Actual); Status verified 2022-11

CONDITIONS: Diabetes Mellitus; Arrhythmias, Cardiac
MeSH Terms: conditions — Diabetes Mellitus; Arrhythmias, Cardiac | interventions — Centrifugation

STUDY DESIGN:
Intervention Model Description: Comparing layperson centrifuge tolerance between diabetics, individuals with past medical history of cardiac arrhythmia, and control subjects. All subjects will participate in the same protocols.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Diabetic Subjects (Other): Individuals with history of diabetes mellitus
  Interventions: Other: Centrifugation
- Subjects with history of arrhythmia (Other): Individuals with history of cardiac arrhythmia
  Interventions: Other: Centrifugation
- Control Subjects (Other): Individuals without history of either Diabetes or cardiac arrhythmia
  Interventions: Other: Centrifugation

INTERVENTIONS:
Other: Centrifugation — Subjects will participate in up to seven different centrifuge profiles over a single day of training (approximately 8 hours). Exposures are design to simulate a spaceflight profile using acceleration anticipated for commercial spaceflights.

SUMMARY:
The study will involve exposing individuals with a known past medical history of diabetes mellitus and/or cardiac arrhythmias to centrifuge-induced acceleration force (G-force) in the NASTAR AFTS-400 simulator to evaluate their response to such forces. Subjects without a history of these conditions will also undergo centrifuge-induced G-forces as controls. This study will contribute to the knowledge of how individuals with such medical conditions experience G-forces that may be experienced during commercial spaceflights.

DETAILED DESCRIPTION:
UTMB has received grant funding from the Federal Aviation Administration (FAA) under the Center of Excellence for Commercial Space Transportation to investigate these topics. The concern is whether spaceflight, an already hazardous endeavor, would be a greater hazard for the less healthy individual. It remains difficult to predict how particular disease processes will respond to the hypergravity environment during launch and landing of spacecraft, and exactly what these hazards may entail.

Conditions such as diabetes mellitus and cardiac arrhythmias may be prevalent in the population group of potential future spaceflight participants and may present additional risk factors in the hypergravity environment, from acceleration tolerance to the ability to carry out moderately complex tasks in emergency or high-stress operational scenarios. While certain disease-related sequelae (such as severe retinopathy, nephropathy, autonomic dysfunction, cardiac ischemia, etc) are likely to represent criteria for exclusion from near-future spaceflight activity, the inclusion of individuals with well-controlled disease without significant sequelae is desirable in the commercial spaceflight industry.

The purpose of this study is to evaluate the tolerance of acceleration forces, induced by centrifuge, in individuals with diabetes mellitus and cardiac arrhythmias. Investigators will include in the study individuals known to have either of the following:

1. Well-controlled diabetes (type I or type II, controlled with diet, oral medications, or insulin injections, with HbA1c of <8% and baseline pre-prandial blood glucose of <250).
2. Well-controlled cardiac arrhythmias (including control via oral medications, implanted pacemakers, or prior ablation or similar intervention). Cardiac arrhythmias of interest include Wolff-Parkinson-White (WPW), atrial fibrillation, atrial flutter, supraventricular tachycardia, accelerated idioventricular rhythms, junctional rhythms, A-V block. Use of an implanted pacemaker, if demonstrated to be successful in controlling prior dysrhythmia, is acceptable.

Investigators will further screen individuals with no known history of these diseases to act as a control group. It is anticipated that individuals with the controlled disease processes included in this study will tolerate acceleration forces well, with changes in cardiovascular responses related primarily to use of medications (primarily beta-blockers; see above for explanation). Investigators will also examine the performance, of both those with medical conditions and the controls, during a simulated emergency with a moderately difficult assigned task. It is hypothesized that these diseases, when well-controlled, are not a contraindication to space travel.

ELIGIBILITY:
Inclusion Criteria:

* We aim to screen individuals known to have either of the following: (1) well-controlled diabetes mellitus (Type I or Type II, controlled with diet, oral medications, or insulin injections or pump) with an HbA1c of <8% or (2) well-controlled cardiac arrhythmias (including control via oral medications, implanted pacemakers, prior ablation or similar intervention). Cardiac arrhythmias of interest include Wolff-Parkinson-White (WPW), atrial fibrillation, atrial flutter, supraventricular tachycardia, accelerated idioventricular rhythms, junctional rhythms, A-V block. Use of an implanted permanent pacemaker (single- or dual-chamber, continuous or demand), if demonstrated to be successful in controlling prior arrhythmia, is acceptable. History of a one-time defibrillation event followed by successful ablation and/or management of an underlying disorder/arrhythmia is acceptable.

Subjects with a history of both diabetes mellitus and cardiac arrhythmia are considered eligible for inclusion if both diseases meet inclusion criteria. The presence of other medical diseases (for example, history of prior myocardial infarction or stenting), if well-controlled, will still be considered eligible for inclusion (see exclusion criteria).

We will further screen individuals with no known history of significant medical disease to act as a control group.

Exclusion Criteria:

* Disease-specific exclusion criteria include:
* Subjects with diabetes:

  * An HbA1c ≥8%
  * Demonstration of poor glucose control (with average preprandial baseline blood glucose of >250)
  * Evidence of advanced disease or sequelae of long-term poor glucose management, such as significant or end-stage renal disease (creatinine of > 3.0 or reliance on hemodialysis), autonomic dysfunction, or diabetic retinopathy
  * "Pre-diabetic" with normal HbA1c (<6.5%), no medications, no lifestyle changes
* Subjects with cardiac arrhythmia:

  * Evidence of symptomatic arrhythmias (for example, frequent light-headedness, syncopal events)
  * Documentation of historical defibrillation events (note that a one-time defibrillation followed by intervention (example: ablation) and complete resolution of arrhythmic activity will NOT be considered exclusionary)
  * Presence of an automated implanted cardiac defibrillator (AICD)
  * History of ventricular tachycardia or ventricular fibrillation, if not otherwise related to an underlying and resolved condition
  * Evidence of cardiac ischemia during any stress testing, severe vascular disease, or similar severe and uncontrolled medical problems identified by any historical documentation or pre-flight screening

Female subjects will be required to be screened for pregnancy; pregnant patients will be excluded from this study. Subjects with extensive experience in the hypergravity environment, such as high performance or acrobatic pilots, will be ineligible.

In addition, significant medical disease other than the diseases of interest may be exclusionary, particularly if they represent identifiable risk previously considered exclusionary from prior hypergravity exposure and centrifuge trials. Examples include:

* Poorly controlled hypertension (baseline systolic >180mmHg, baseline diastolic >100 mmHg)
* History of cardiac transplant
* History of cardiac ejection fraction of <50%
* Lung disease or cardiac disease requiring continuous supplemental oxygen therapy
* Acute spinal/neck/back injury
* Acute post-surgical period (<6wks)
* Severe obesity, with weight >250lbs
* History of unpredictable or uncontrollable psychiatric outbursts, disruptive behavior, etc

Participants with significant cardiac risk factors beyond age and sex (including a history of tobacco use, a history of hyperlipidemia or dyslipidemia, a history of hypertension or blood pressure management with medication, or a history of diabetes) will be required to provide further information including lipid panels, HbA1c in the case of diabetes, and exercise stress testing. Patients will be excluded for:

* Evidence of cardiac ischemia during stress testing, with examples including:

  * exercise-induced angina
  * exercise-induced hypotension
  * evidence of ≥1mm electrocardiogram ST-segment depression induced by exercise or pharmacological stress
  * reversible ischemia on myocardial perfusion imaging
* Severe coronary vascular disease, with examples including:

  * evidence of reversible ischemia on myocardial perfusion imaging,
  * known history of multi-vessel coronary artery disease that has not received stenting or surgical correction (or is not amenable to stenting or surgical correction)
* Similar severe and uncontrolled medical problems identified by any of the screening medical monitors or physicians.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-09-27 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Heart Rate | 5 seconds after the onset of acceleration
  Abnormalities of heart rate (bpm) including bradycardia (<55bpm) or tachycardia outside of expected norms (>180) during acceleration phases
Systolic Blood Pressure - before | 5 minutes before centrifuge profile
  Measurement of systolic blood pressure (mmHg) at 5 minutes prior to centrifuge profile
Diastolic Blood Pressure - before | 5 minutes before centrifuge profile
  Measurement of diastolic blood pressure (mmHg) at 5 minutes prior to centrifuge profile
Systolic Blood Pressure - after | 5 minutes before centrifuge profile
  Measurement of systolic blood pressure (mmHg) at 5 minutes after centrifuge profile
Diastolic Blood Pressure - after | 5 minutes after centrifuge profile
  Measurement of diastolic blood pressure (mmHg) at 5 minutes after centrifuge profile
Blood Glucose | continuous blood glucose monitoring for 8 hours during day of testing
  Blood glucose (g/dL) range on the day of testing
ECG dysrthythmias | up to 12 min, assessed during the duration of acceleration exposure
  Presence of dysrhythmias including PACs, PVCs, AIVR, or other rhythm alterations
Errors during Emergency Scenario | approximately 1 min, immediately following final acceleration profile
  During a simulated Emergency, subjects will enter 12 keystrokes on a touch-screen interface following completion of acceleration profiles. Outcome measures will include number of entry errors (e.g. wrong button, wrong order) during this examination
Time of data entry completion during Emergency Scenario | approximately 1 min, immediately following final acceleration profile
  During a simulated Emergency, subjects will enter 12 keystrokes on a touch-screen interface following completion of acceleration profiles. Outcome measures will include the time to completion of all 12 keystrokes.

CONTACTS AND LOCATIONS:
Overall Officials: William Powers, MD, Principal Investigator — The University of Texas Medical Branch, Galveston
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No